CLINICAL TRIAL: NCT01089738
Title: An Investigator And Subject-blind Phase 1 Study To Characterize The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Doses Of Pf-03382792 In Healthy Elderly Subjects
Brief Title: A Study To Look At Safety And Blood Concentrations After Multiple Doses Of PF-03382792 In Healthy Elderly Individuals
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: B1651003
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: mulitple dose; pharmacokinetics; safety; healthy elderly volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dosing (Experimental): Ascending Doses
  Interventions: Drug: PF-03382792 0.5mg; Drug: PF-03382792 1.5 mg; Drug: PF-03382792 5 mg; Drug: PF-03382792 15 mg

INTERVENTIONS:
Drug: PF-03382792 0.5mg — 0.5 mg PF-03382792, qd, for 14 days or placebo
Drug: PF-03382792 1.5 mg — 1.5 mg PF-03382792, qd, for 14 days or placebo
Drug: PF-03382792 5 mg — 5 mg PF-03382792, qd, for 14 days or placebo
Drug: PF-03382792 15 mg — 15 mg PF-03382792, qd, for 14 days or placebo

SUMMARY:
This study is designed to look at the safety and blood concentrations of PF-03382792 in healthy elderly subjects after taking multiple doses for 14 days.

DETAILED DESCRIPTION:
To examine safety, toleratibilty and pharmacokinetics of PF-03382792 in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged 65-80 years old
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2
* Total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subjects with symptoms or signs of adrenal insufficiency.
* Subjects with clinically significant ocular lens abnormalities as detected by the investigator based on the findings of a slit lamp examination performed by an ophthalmologist.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2011-04-25 (Estimated); Study Completion 2011-04-25 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoints include: AEs, vital signs, triplicate ECGs, | Day 0 to Day 28
Safety Endpoints include: Cosyntropin Stimulation Test, Clinical Examinations, Slit Lamp Examination, Aldosterone Concentrations | Day 0 to Day 28
Safety Endpoints include: safety laboratory endpoints (including a complete blood count and a full chemistry panel, including electrolytes, hepatic transaminases, and urinalysis, with microscopic analysis if dipstick analysis is positive), | Day 0 to Day 28
Pharmacokinetic endpoints include: Plasma concentrations of PF 03382792 and its N dealkylated metabolite, PF 03227077, will be measured and used to determine Cmax, Tmax, AUC on Day 1 and Css,max, Tss,max, AUC, Css,min, Css,avg on Days 7 and 14. | Day 0 to Day 28
Additional pharmacokinetic endpoints: the accumulation ratio (Rac) will be determined from Day 14 and Day 1 AUC. If data permit, t1/2 and urinary excretion parameters (CLR for the parent and Ae and Ae%) will be calculated. | Day 0 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1651003&StudyName=A%20Study%20To%20Look%20At%20Safety%20And%20Blood%20Concentrations%20After%20Multiple%20Doses%20Of%20PF-03382792%20In%20Healthy%20Elderly%20Individuals%0A